CLINICAL TRIAL: NCT05428943
Title: A Phase 1b Study of OPT101 in Patients With Type 1 Diabetes
Brief Title: OPT101 in Type 1 Diabetes Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Op-T LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OPT101-100-20
Record Dates: First submitted 2022-06-09; First posted 2022-06-23 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OPT101 1.1 mg/kg and Placebo (Other): 9 subjects (6 investigational product:3 placebo)
  Interventions: Drug: OPT101
- OPT101 2.8 mg/kg and Placebo (Other): 9 subjects (6 investigational product:3 placebo)
  Interventions: Drug: OPT101

INTERVENTIONS:
Drug: OPT101 — 15-mer peptide derived from the sequence of mouse CD154.

SUMMARY:
Phase 1b designed to assess safety, pharmacokinetics, immunological and clinical effects of multiple ascending doses of OPT101.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give informed consent for the trial
2. Male or female aged ≥18 years on the day of signing informed consent
3. Diagnosis of Type 1 diabetes (T1D) within the last 20 years
4. Is medically stable based on physical examination, medical history, laboratory results, and vital signs performed at screening
5. Women of childbearing potential must have a negative highly sensitive serum test (beta-human chorionic gonadotropin) at screening and a negative urine pregnancy test at the Visit 1 Day 1 prior to receiving the investigational product.
6. Women must agree to use one of the following methods of birth control for the duration of the clinical trial: systemic hormonal contraceptive (oral, injected, transdermal), intrauterine device, double barrier (e.g., cervical cap or diaphragm with condom or spermicide). Men with female partners must agree to use double barrier contraception, unless their partner is using systemic hormonal contraceptives or has an intrauterine device.

   -

Exclusion Criteria:

1. Is over the age of 60 years old
2. Currently has or had a history of malignancy
3. Has an immune deficiency syndrome (for example, severe combined immunodeficiency syndrome, T-cell deficiency syndromes, B-cell deficiency syndromes, or chronic granulomatous disease), or bone marrow or organ transplantation, or a disease associated with lymphopenia
4. Is currently receiving an immuno-modulatory treatment.
5. Patients with a history of venous and arterial thromboembolic events including, but not limited to, the following: deep venous thrombosis, pulmonary embolism, myocardial infarction, stroke, transient ischemic attack, or arterial insufficiency causing digital gangrene should be excluded. In addition, patients with recent immobilization or recent surgery, should be excluded. Patients with a history of abnormal prothrombotic laboratories such as congenital or inherited deficiency of antithrombin III, protein C, protein S, or confirmed diagnosis of antiphospholipid syndrome should also be excluded.
6. Has active infections, is prone to infections or has chronic, recurrent or opportunistic infectious disease, including but not limited to, Epstein-Barr virus (EBV), cytomegalovirus (CMV) chronic renal infection, chronic chest infection, sinusitis, recurrent urinary tract infection, Pneumocystis carinii, aspergillosis, latent or active granulomatous infection, histoplasmosis, or coccidioidomycosis or an open, draining, or infected non-healing skin wound or ulcer
7. Has recent or active hepatitis A infection, current/chronic hepatitis B and hepatitis C infection, or HIV infection. Participants with immunity to hepatitis B from previous infection (defined as negative HBsAg, positive anti-HBc, and positive hepatitis B surface antibody [anti-HBs]) or vaccination (defined as negative HBsAg, negative anti-HBc, and positive anti-HBs) may be eligible to participate.
8. Has a history of latent or active TB
9. Has received a live (attenuated) vaccine within the last 60 days, including patients who plan to receive live (attenuated) vaccines during the study or within 60 days after the final dose of study treatment.
10. Patients with clinically significant abnormal laboratory test values in screening blood samples. In particular patients with the following should be excluded:

    i. Patients with abnormal coagulation panel at screening such as abnormal PT or aPTT or fibrinogen ii. Abnormal liver function tests:

1. Liver enzyme abnormalities (except in the case of known Gilbert's syndrome) 2. AST or ALT ≥3x ULN and total bilirubin ≥2x ULN 3. AST or ALT ≥5x ULN 4. AST or ALT ≥3x ULN if associated with appearance or worsening of rash or hepatitis symptoms iii. Abnormal platelet counts (<150,000mcL or > 450,000mcL) iv. Abnormal white blood cell counts (<3mL or > 11mL) v. Abnormal eGFR (<50mg/dL or >1.10mg/dL) vi. Abnormal Factor VIII (> 160%) vii. Abnormal D-Dimer (> 500ng/mL FEU) 11. Patients planning to undergo elective procedures or surgeries at any time after signing the ICF through the follow-up visit.

12. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

13. Recent history of bleeding or bleeding disorders or any condition whereby in the opinion of the treating investigator giving anti-coagulation during treatment would be contraindicated.

14. History of hypersensitivity to antihistamines. 15. Weight is over 250lbs. 16. Patients with active drug or alcohol abuse within 1 year prior to screening 17. Patient is participating in a clinical trial of another investigational drug or device, including patients who have participated in another study for a duration of 5 half-lives of the investigational agent.

18. Patient is a prisoner 19. Investigators could exclude patients with any medical condition, including, but not limited to, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal, or a psychiatric condition that, in the opinion of the Investigator, could compromise the participant's ability to participate in this study.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 90 days
  Treatment related adverse events will be recorded and assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Serum samples collected to determine AUC0-t | 90 days
  Blood samples will be collected to determine the serum concentrations of OPT101 (mg/kg)
Serum samples collected to determine Cmax | 90 days
  Blood samples will be collected to determine the serum concentrations of OPT101 (mg/kg)
Serum samples collected to determine CL/F | 90 days
  Blood samples will be collected to determine the serum concentrations of OPT101 (mg/kg)
Serum samples collected to determine t1/2 | 90 days
  Blood samples will be collected to determine the serum concentrations of OPT101 (mg/kg)
Serum samples collected to determine HbA1C from baseline pre mixed meal tolerance test | 90 days
Serum samples collected to determine c-peptide post mixed meal tolerance test | 90 days
Serum samples collected to determine glucose levels (mmol/L) pre and post mixed meal tolerance test | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Boswell, MS, Study Director — OP-T
Locations (2):
- United States (2):
  - Diablo Clinical Research Center, Walnut Creek, California
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No